CLINICAL TRIAL: NCT03096522
Title: A Randomized Controlled Trial on the Effect of Topical Phenytoin 2% on Wound Healing After Fistulotomy
Brief Title: Randomized Trial on the Effect of Topical Phenytoin on Healing After Fistulotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mansoura33
Record Dates: First submitted 2017-03-26; First posted 2017-03-30 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula | interventions — Phenytoin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenytoin 2% spray (Active Comparator): Patients undergoing anal fistulotomy with postoperative topical phenytoin therapy
  Interventions: Drug: Phenytoin 2% spray; Procedure: Anal fistulotomy
- Anal fistulotomy (Active Comparator): Patients undergoing anal fistulotomy without postoperative topical therapy
  Interventions: Procedure: Anal fistulotomy

INTERVENTIONS:
Drug: Phenytoin 2% spray — Patients will undergo anal fistulotomy then they will use phenytoin 2% spray topically on the anal wound resulting from fistulotomy with each sitz bath (twice per day) untill the anal wound heals completely
  Other Names: Healosol
  Arms: Phenytoin 2% spray
Procedure: Anal fistulotomy — Probing of the fistula tract followed by lay open of the tract and curettage of granulation tissue in its base
  Other Names: Lay open of anal fistula tract

SUMMARY:
Patients with anal fistula who will undergo anal fistulotomy will be randomized into one of two groups; the first group will receive topical phenytoin therapy postoperatively and the second group will not receive such topical treatment.

DETAILED DESCRIPTION:
Patients with anal fistula who will undergo anal fistulotomy will be randomized into one of two groups; the first group will receive topical phenytoin therapy postoperatively and the second group will not receive such topical treatment.

Healing of the wound after fistulotomy will be observed every week and the duration till complete healing will be recorded. The two groups will be compared regarding the mean duration till complete healing and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aging between 18-65 years with primary simple anal fistula (subcutaneous, intersphincteric, or low trans-sphicnteric involving less than 25% of external anal sphincter fibers)

Exclusion Criteria:

* Patients with high trans-sphincteric, extra-sphincteric, supra-sphincteric, secondary, or recurrent anal fistulas.
* Patients with associated anorectal pathology such as anal fissure, hemorrhoids, rectal prolapse, neoplasm, solitary rectal ulcer, and inflammatory bowel diseases.
* Patients under chronic corticosteriod or immunosuppressive therapy.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
Healing | 4-8 weeks
  Complete epithelilization of the fistulotomy wound without persistent external openings or discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D., Principal Investigator — Mansoura University, Faculty of medicine
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No